CLINICAL TRIAL: NCT05980585
Title: Assessment of Heart Failure (HF) At-Home Management Solution ADI Cardio Pulmonary Monitoring System (CPM)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Analog Device, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OBS-BAPTISTJAX
Record Dates: First submitted 2023-07-26; First posted 2023-08-08 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: The study looks at a single group of patients that uses the CPM Device
Masking Description: The participant, the investigator, and the outcomes assessor will all be masked to the device data during the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Study Group (Experimental): The Study group will use the CPM device once daily (in the morning) for 60 days.
  Interventions: Device: CPM Device

INTERVENTIONS:
Device: CPM Device — Daily use of the CPM wearable device

SUMMARY:
This study is meant primarily to assess the deployment of the ADI CPM System in a clinical setting and determine interoperability of the CPM System within existing care pathways for patients with CHF. In this initial study the CPM System will not be used to determine or support clinical decision making however post deployment the clinical study team will review patient HF events and changes in treatment during the course of the deployment and compare to the data generated by the CPM System during the study to determine the accuracy of the patient generated data as a basis for designing a more comprehensive "interventional study" to determine clinical and financial efficacy of the CPM System.

DETAILED DESCRIPTION:
Patients will be recruited and begin the study as they are identified and consent to the study. Recruiting will end either by a designated date set at the initiation of the study or when 30 patients have been enrolled in the study.

The duration of the study for each patient will be approximately 60 days beginning with the baseline/initial visit and concluding 30 days after the patient has completed device use. The patient will use the device given to the once a day during the first 60 days the study and following that time patient records will be reviewed retrospectively for CHF events for the 60 days plus an additional 30 days after their last measurement. Each patient will also receive weekly calls from the research team to check in on device functionality and assure adherence to the protocol.

At visit 1, the start of the study, baseline information will be collected, importantly including accurate weight and notes about congestion and fluid buildup. The study will be re-described to the participant. The research team will then set up the device for the individual patient by making adjustments (as needed) to address patient specific anatomy), ensuring that the sensors are all contacting the appropriate chest areas, and confirming the measurements on the CPM Web application. The patient will be shown how to apply and replace the adhesive on the device, how to position the device, how to take a measurement with the device, and how to store the device on the Base Station. The trained provider will then register the baseline reading for the CHF device using the CHF Mobile App.

Informational materials about using the device, refreshing adhesives, and meanings of LEDs and chimes on the device will also be given to the patient. The patient will be instructed to follow the normal regimen prescribed by their by their physician, but to add taking a measurement with their CPM at the same time each day (preferably when they first wake up).

Between visits, caregivers will not have any access to the data being collected on the CHF Device. They should perform their usual standard of care on these patients. Participants will also receive calls from the research team to check in about the progress of the study (i.e., if protocols are being followed correctly, if the CPM device is working properly, and if adherence is satisfactory. This check-in, conversation topics should focus on any ease-of-use issues and address any compliance-based issues.

The ADI team will have access to data (without any patient identifying information) throughout the course of the trial, including adherence rates of patients. The sponsors will reach out to the study team if a specific patient is found to have missed 2 days in a row of measurements. The research team will contact patients directly if there is a continued trend towards non-compliance.

If a participant is having technical difficulties using the CPM System, the research team in conjunction with ADI will provide direct (in office) or remote assistance or replace existing equipment as necessary.

On visit 2, which will take place at the end of the 60 days, the research team will make arrangements for the patient to return to the office for a check-up and return the device (the same tests as described in the "physical examination" section including b lines/comet tails, dyspnea scale, etc.). Patients will also be asked about their perception on "ease of use", impact on day-to-day activities, and overall satisfaction with the CPM system. Thirty days following the last measurement the study team, will review the patients records for all HF related events and treatment changes.

ELIGIBILITY:
Inclusion Criteria: one or more of the following

* NYHA Class III-IV HF
* NYHA Class II HF patients with elevated BNP levels (BNP>100 pg per mL) NYHA Class II HF patients with elevated NT-proBNP levels (NT-proBNP>400 pg per mL)
* HF Patients with at least one Worsening HF event (in /out-patient) in past 12 months
* HF patients with Acute Renal Failure or Chronic Kidney Disease
* HF patients with Chronic Obstructive Pulmonary Disease (COPD)
* HF patients currently on 40 mg or more of Furosemide /

Exclusion Criteria:

* Under age 60
* End Stage Renal Disease
* Patients with severe COPD (GOLD stage III or IV)
* Limited mobility preventing application of device
* Cognitive impairments that would limit the application and proper use of the device
* Skin allergies or skin sensitivities to silicone-based adhesives
* Pregnancy
* Skin breakdown on the left chest or breast area
* Not willing to shave chest hair if needed to apply device
* No cellular coverage (Patient's Home)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-20 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Interoperability of CPM system | 60 days
  patient satisfaction with system obtained through survey questions; ease of use, impact and satisfaction; scale of 1-7 used with 1 being negative and 7 being positive, impact on daily life obtained though Minnesota Living with Heart Failure questionnaire

SECONDARY OUTCOMES:
Correlation of device data and clinical outcomes | 90 days
  Retrospective review of data to determine correlation of patient specific device measurements (such as increase/decrease in specific device parameters) with heart failure events. Measurements include thoracic impedance, respiration rate (RR), heart rate (HR), relative tidal volume (rTV), RR variability, HR variability, RR/rTV, QRS width, QTc width, presence of atrial fibrillation, and diastolic heart sound strength

CONTACTS AND LOCATIONS:
Locations (1):
- Baptist Health, Jacksonville Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No